CLINICAL TRIAL: NCT01894308
Title: A Multiple-Dose, Single Period, Phase II Dose Ranging Study to Examine TDS-Testosterone 5% in Adult Male Subjects
Brief Title: A Dose Ranging Study to Examine TDS-Testosterone 5%
Acronym: PARC-T-D
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Transdermal Delivery Solutions Corp (Industry)
Collaborators: Advanced Therapies Centre, The London Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARC-Testosterone-D1/09/13; 2013-001766-42 (EudraCT Number); IRAS project ID: 146877 (Other: NHS London - West London & GTAC Research Ethics Committee)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Hypogonadotropism
Keywords: Male Hormone Replacement; Multiple Dose; Single Period; Phase II; Dose Ranging; Adult Male Subjects; Testosterone Replacement
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Forearm dose (Active Comparator): Half of Ss will receive their dose of Testosterone on the inner aspects of their forearms.
  Interventions: Drug: Testosterone; Device: Pump Sprayer
- Chest Dose (Active Comparator): Half of Ss will receive their dose of Testosterone on the chest.
  Interventions: Drug: Testosterone; Device: Pump Sprayer

INTERVENTIONS:
Drug: Testosterone — 10,30,50 and 70 mg doses of micronized Testosterone delivered by means of a new liquid transdermal delivery solution, HypoSpray(R)once daily for 7 days or until halted due to systemic or dermal reactions.
Device: Pump Sprayer — A dose of product solution is delivered by means of a metered pump spray.

SUMMARY:
This study is a continuation of previous studies done in healthy volunteers to prove the efficacy of delivering Testosterone, the male hormone, rapidly across intact skin in s series of doses from low to high in men with low-to-no natural testosterone production to measure their response to the varying doses. The results of this study will inform further studies which will be longer in length, as to the starting doses. The study will be conducted in London, U.K. at the Advanced Therapies Centre, The London Clinic.

DETAILED DESCRIPTION:
48 Patients will be enrolled following 2 independent verifying blood tests of their diagnosis of Hypogonadism. there will be 4 cohorts of 12 subjects, each receiving doses of the trail materials, titrated by means of number of sprays applied. Doses will range from 10 to 70 mgs Testosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Hypogonadal Male subjects - morning testosterone level ≤300 ng/dL (10.4 ng/L).
2. 18 and 75 years of age, inclusive.
3. The subject is willing and able to read, understand the Subject Information Sheet and provide written informed consent.
4. The subject has a body mass index (BMI) within 18-30 kg/m2.
5. The subject is in otherwise good health as determined by medical history and physical examination.
6. The subject is a non-smoker.
7. The subject must agree to comply with the placement of an indwelling catheter on two separate occasions and the drawing of blood samples for the pharmacokinetic assessments.
8. The subject is willing and able to comply with all testing and requirements defined in the protocol.
9. The subject is willing and able to return to the study site for all visits.

Exclusion Criteria:

1. The subject has any relevant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator, particularly an elevated PSA reading >4.0 ng/ml or ALT and AST greater than 2 times the upper limit of normal, clinically significant anemia (hematocrit <35%) or renal dysfunction (creatinine >2mg/dL), active deep vein thrombosis, thromboembolic disorders or history of these conditions.
2. The subject has had a clinically significant illness within 30 days preceding entry into this study.
3. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
4. The subject has a known allergy or history of hypersensitivity to Testosterone or similar compounds.
5. The subject has used any prescription medication within 14 days or over-the-counter (OTC) medication or alcohol within 48 hours of dosing or intends to use any prescription or OTC medication during the study that may interfere with the evaluation of study medication.
6. The subject has donated or lost a significant volume of blood (>450 mL) within four (4) weeks of the study, and their haemoglobin concentration and haematocrit have not returned to within 5% of normal.
7. The subject has a Hematocrit level > 51%
8. The subject has a history of substance abuse or a current positive urine drug screen or urine alcohol test.
9. Alcohol consumption greater than community norms (i.e. more than 21 standard drinks per week for males).
10. Subjects who have received an investigational drug or have used an investigational device in the 30 days prior to study entry.
11. Subjects with an American Urological Association System Index for Prostatism score greater than 7
12. Subjects with a history of prostate or breast carcinoma.
13. Subjects with prostatic mass on screening physical examination.
14. Subjects with a history of significant skin disease.
15. Subjects with a history of sleep apnea.
16. Subject with a partner with a history of breast cancer.
17. Subject with a partner of child bearing potential who is not willing to use adequate contraception for the duration of the trial.
18. Subject whose partner is pregnant.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Dose Range Measure of serum levels of testosterone in response to varying doses | 1 week
  A pharmacokinetic measure of serum levels of testosterone in response to varying doses of from 10 to 70 mgs of Testosterone.

SECONDARY OUTCOMES:
Dermal Safety as measured by | 1 Week
  Incidence of treatment-emergent side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Shern L. Chew, M.D., Ph.D., Principal Investigator — Consultant Physician and Professor of Endocrine Medicine
Locations (1):
- Advanced Therapies Centre, The London Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chik Z, Johnston A, Tucker AT, Chew SL, Michaels L, Alam CA. Pharmacokinetics of a new testosterone transdermal delivery system, TDS-testosterone in healthy males. Br J Clin Pharmacol. 2006 Mar;61(3):275-9. doi: 10.1111/j.1365-2125.2005.02542.x. PMID 16487220